CLINICAL TRIAL: NCT02501863
Title: Analgesic Effect of Ropivacaine Plus Fentanyl vs Ropivacaine for Continuous 3-in-1 FNB After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Center, Seoul (Other)
Responsible Party: Principal Investigator, Mija Yun, MD, PhD, Anesthesiologist, National Medical Center, Seoul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN1
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine+fentanyl (Experimental): Femoral nerve block with ropivacaine+fentanyl
  Interventions: Femoral nerve catheter insertion, spinal anesthesia, IV-PCA with hydromorphone.
  Interventions: Drug: Femoral nerve block with ropivacaine+fentanyl
- Ropivacaine (Experimental): Femoral nerve block with ropivacaine
  Interventions: Femoral nerve catheter insertion, spinal anesthesia, IV-PCA with hydromorphone.
  Interventions: Drug: Femoral nerve block with ropivacaine

INTERVENTIONS:
Drug: Femoral nerve block with ropivacaine+fentanyl — Ropivacaine+fentanyl are used for continuous femoral nerve block, spinal anesthesia, IV-PCA with hydromorphone
  Other Names: RF
  Arms: Ropivacaine+fentanyl
Drug: Femoral nerve block with ropivacaine — Ropivacaine is used for continuous femoral nerve block, spinal anesthesia, IV-PCA with hydromorphone
  Other Names: R
  Arms: Ropivacaine

SUMMARY:
The postoperative analgesic effect of the continuous 3-in-1 femoral nerve block (FNB) with ropivacaine/fentanyl or with ropivacaine were compared in total knee arthroplasty.

DETAILED DESCRIPTION:
Forty patients of American Society of Anesthesiologist physical status Ⅰor Ⅱ undergoing total knee arthroplasty under spinal anesthesia would be enrolled and randomly divided into two groups (R, "3-in-1" using a 30 ml of ropivacaine 0.375% and a continuous 3-in-1 with a ropivacaine 0.2%(8mL/h) for 48 h after operation, RF: Fifty ug of fentanyl will be added to a bolus(30ml ropivacaine 0.375%) and 1ug/ml of fentanyl will be mixed to a continuous infusion(8mg/h, ropivacaine 0.2%). Spinal anesthesia will be done after the insertion of femoral catheter. IV PCA with hydromorphone(0.15mg/ml, 0-1-10), will be used for rescue analgesics. Visual analgesia scale, hydromorphone consumption, side effects until 48h after operation and satisfaction will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1 to 3 undergoing total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* Patients were excluded from this study if they had contraindications to a regional anesthetic technique (e. g., local infection, sepsis, coagulation abnormality), allergy to local anesthetic or fentanyl, preexisting neurologic deficit in the lower extremities, and inability to comprehend the pain scales or use IV patient-controlled analgesia (PCA) device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain on the VAS(Visual Analog Scale) | During 48 hour after operation
  VAS(resting, movement) at operation day, postoperation 1 day, postoperation 2 day.

SECONDARY OUTCOMES:
Number of participant with side effects | During 48 hour after operation

CONTACTS AND LOCATIONS:
Overall Officials: Mijung Yun, MD, PhD, Principal Investigator — National medical center

IPD SHARING:
Plan to Share IPD: No